CLINICAL TRIAL: NCT05233280
Title: Early Versus Delayed Oral Liquids and Soft Food After Elective Ceasarean Section
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: Oral feeding after ceasarean
Record Dates: First submitted 2022-01-01; First posted 2022-02-10 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2021-12

CONDITIONS: Prevent Postopertive Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — Fluid Therapy; Postoperative Period

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Early feeding group
  Interventions: Other: Oral liquids and soft food 2 hours postoperative
- Group B: Delayed feeding group

INTERVENTIONS:
Other: Oral liquids and soft food 2 hours postoperative — Early versus delayed oral liquid feeding after ceasarean section
  Groups: Group A

SUMMARY:
To compare the safety of early versus delayed oral feeding after uncomplicated cesarean section under spinal anesthesia

DETAILED DESCRIPTION:
Cesarean section is one of most common surgical procedures saving both for mother and newborn when medically indicated .traditionally patients are not given fluids or food afer abdominal surgery until bowel function return as evidenced by bowel sounds passage of flatus or stool or feeling of hunger the rationale of this practice is to prevent postoperative nausea , vomiting, distension and other complications

ELIGIBILITY:
Inclusion Criteria:

* previous 1,2,3 cs Uncomplicated elective cs Singletone pregnancy Spinal anesthesia

Exclusion Criteria:

* women with medical disorder HTN, DM History of bowel surgery or intraoprative complication Contraindication to spinal anesthesia

Ages: 17 Years to 50 Years | Sex: Female
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Women in child bearing period
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-02-20 (Estimated); Primary Completion 2022-03-15 (Estimated); Study Completion 2022-04-15 (Estimated)

PRIMARY OUTCOMES:
Time of passage of flatus | 6 hrs